CLINICAL TRIAL: NCT03414983
Title: An Open-Label Exploratory Phase 2/3 Study of Nivolumab With Standard of Care Therapy vs Standard of Care Therapy for First-Line Treatment of Metastatic Colorectal Cancer
Brief Title: An Investigational Immunotherapy Study of Nivolumab With Standard of Care Therapy vs Standard of Care Therapy for First-Line Treatment of Colorectal Cancer That Has Spread
Acronym: CheckMate 9X8
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9X8; 2017-003662-27 (EudraCT Number)
Record Dates: First submitted 2018-01-24; First posted 2018-01-30 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Nivo + SOC
  Interventions: Biological: Nivolumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Bevacizumab
- Arm B (Active Comparator): SOC
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Bevacizumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Arm A
Drug: Oxaliplatin — Specified dose on specified days
Drug: Leucovorin — Specified dose on specified days
  Other Names: Calcium Folinate
Drug: Fluorouracil — Specified dose on specified days
Drug: Bevacizumab — Specified dose on specified days
  Other Names: Avastin

SUMMARY:
This purpose of this study is to evaluate nivolumab (BMS-936558) in combination with standard of care (SOC) chemotherapy with bevacizumab for the treatment of first-line metastatic colorectal cancer (mCRC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal cancer, not amenable to curative resection
* No prior chemotherapy for metastatic colorectal cancer
* ECOG Performance Status of 0-1
* Ability to provide adequate tissue sample

Exclusion Criteria:

* Patients with clinically relevant medical history, including autoimmune disease, cardiovascular disease, hepatic disease or bleeding disorders
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Suibb
Locations (49):
- United States (35):
  - Uab Comprehensive Cancer Center, Birmingham, Alabama
  - Local Institution - 0004, Los Angeles, California
  - Local Institution - 0010, Aurora, Colorado
  - Local Institution - 0027, Denver, Colorado
  - Local Institution - 0020, New Haven, Connecticut
  - Local Institution - 0039, Miami, Florida
  - Local Institution - 0047, St. Petersburg, Florida
  - Local Institution - 0033, Arlington Heights, Illinois
  - Local Institution - 0044, Indianapolis, Indiana
  - Local Institution - 0021, Bethesda, Maryland
  - Local Institution - 0003, Boston, Massachusetts
  - Local Institution - 0049, Boston, Massachusetts
  - Local Institution - 0052, Boston, Massachusetts
  - Local Institution - 0053, Boston, Massachusetts
  - Local Institution - 0035, Minneapolis, Minnesota
  - Local Institution - 0002, Rochester, Minnesota
  - Local Institution - 0032, Papillion, Nebraska
  - Local Institution - 0029, Henderson, Nevada
  - Local Institution - 0031, Johnson City, New York
  - Local Institution - 0046, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Local Institution - 0038, Portland, Oregon
  - Local Institution - 0005, Philadelphia, Pennsylvania
  - Local Institution - 0024, Pittsburgh, Pennsylvania
  - Local Institution - 0023, Sioux Falls, South Dakota
  - Erlanger Oncology & Hematology - Univ. of TN, Chattanooga, Tennessee
  - Local Institution - 0019, Nashville, Tennessee
  - Local Institution - 0026, Bedford, Texas
  - Local Institution - 0034, Dallas, Texas
  - Local Institution - 0037, Fort Worth, Texas
  - Local Institution - 0040, San Antonio, Texas
  - Local Institution - 0036, Tyler, Texas
  - Local Institution - 0025, Richmond, Virginia
  - Local Institution - 0028, Roanoke, Virginia
  - Local Institution - 0006, Madison, Wisconsin
- Canada (7):
  - Local Institution - 0017, Edmonton, Alberta
  - Local Institution - 0015, Ottawa, Ontario
  - Local Institution - 0014, Toronto, Ontario
  - Local Institution - 0048, Montreal, Quebec
  - Local Institution - 0012, Québec, Quebec
  - Local Institution - 0013, Sherbrooke, Quebec
  - Local Institution - 0016, Trois-Rivières, Quebec
- Japan (3):
  - Local Institution - 0055, Nagoya, Aichi-ken
  - Local Institution - 0051, Kashiwa-shi, Chiba
  - Local Institution - 0050, Sunto-gun, Shizuoka
- Local Institution - 0009, San Juan, Puerto Rico
- Spain (3):
  - Local Institution - 0043, Barcelona
  - Local Institution - 0042, Madrid
  - Local Institution - 0041, Majadahonda - Madrid

REFERENCES:
- [Derived] Lenz HJ, Parikh A, Spigel DR, Cohn AL, Yoshino T, Kochenderfer M, Elez E, Shao SH, Deming D, Holdridge R, Larson T, Chen E, Mahipal A, Ucar A, Cullen D, Baskin-Bey E, Kang T, Hammell AB, Yao J, Tabernero J. Modified FOLFOX6 plus bevacizumab with and without nivolumab for first-line treatment of metastatic colorectal cancer: phase 2 results from the CheckMate 9X8 randomized clinical trial. J Immunother Cancer. 2024 Mar 13;12(3):e008409. doi: 10.1136/jitc-2023-008409. PMID 38485190
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: NIV+mFOLFOX+BEV: Nivolumab 240 mg + Standard of Care (SOC) mFOLFOX6/bevacizuma every 2 weeks
- Arm B: mFOLFOX+BEV: mFOLFOX6/bevacizumab (SOC) every 2 weeks
Period: Pre-Treatment
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Started (Started=Randomized) | 127 | 68
Completed (Completed=Treated) | 123 | 62
Not Completed | 4 | 6
Not completed — Other reasons | 1 | 0
Not completed — Participant no longer meets study criteria | 2 | 3
Not completed — Participant withdrew consent | 1 | 3
Period: Treatment
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Started (Started=Treated) | 123 | 62
Completed | 9 | 0
Not Completed | 114 | 62
Not completed — Participant withdrew consent | 4 | 3
Not completed — Participant request to discontinue study treatment | 8 | 10
Not completed — Adverse Event Unrelated to Study Drug | 5 | 2
Not completed — Death | 0 | 1
Not completed — Study Drug Toxicity | 10 | 5
Not completed — Disease Progression | 75 | 29
Not completed — Not reported | 1 | 0
Not completed — Other reasons | 3 | 2
Not completed — Poor/non-compliance | 2 | 0
Not completed — Maximum clinical benefit | 5 | 9
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative reasons by sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV | Total
Number analyzed (Participants) | 127 | 68 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (13.3) | 57.2 (11.4) | 56.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 19 | 76
  Male | 70 | 49 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 108 | 53 | 161
  Unknown or Not Reported | 12 | 6 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 96 | 57 | 153
  Black or African American | 8 | 2 | 10
  Asian | 15 | 5 | 20
  Other | 6 | 3 | 9
  Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Blinded Independent Central Review (BICR)
Description: Progression Free Survival (PFS) is defined as the time from randomization to the date of the first documented progression, as determined by BICR (per RECIST 1.1), or death due to any cause, whichever occurs first. Baseline tumor assessment is defined as tumor scans prior to or on randomization date. Participants who did not have documented progression per BICR and who did not die or participants who started any subsequent anti-cancer therapy without a prior reported progression per BICR will be censored at the date of the last tumor assessment on or prior to initiation of the subsequent anticancer therapy, if any. Participants who die without a reported prior progression per BICR will be considered to have progressed on the date of death. Participants who did not have any baseline or post baseline tumor assessments and did not die (or died after initiation of the subsequent anti-cancer therapy) will be censored at the randomization date.
Time Frame: From randomization to up to the date of the first documented progression (up to 16 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Months | 11.86 [8.94 to 15.70] | 11.93 [10.09 to 12.19]
Statistical Analysis 1: Comparison: Arm A: NIV+mFOLFOX+BEV vs Arm B: mFOLFOX+BEV; Hazard Ratio is Arm A: NIV+mFOLFOX+BEV over Arm B: mFOLFOX+BEV; Test type: Superiority; p = 0.3022, Log Rank — Stratified regular log-rank test; Hazard Ratio (HR) = 0.81, 80% CI 2-sided [0.61 to 1.07] — Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm A: NIV+mFOLFOX+BEV vs Arm B: mFOLFOX+BEV; Hazard Ratio is Arm A: NIV+mFOLFOX+BEV over Arm B: mFOLFOX+BEV; Test type: Superiority; p = 0.3022, Log Rank — Stratified regular log-rank test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.53 to 1.23] — Stratified Cox proportional hazard model

2. Secondary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: Progression Free Survival (PFS) is defined as the time from randomization to the date of the first documented progression, as determined by Investigator Assessment, or death due to any cause, whichever occurs first. Baseline tumor assessment is defined as tumor scans prior to or on randomization date. Participants who did not have documented progression per Investigator Assessment and who did not die or participants who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the date of the last tumor assessment on or prior to initiation of the subsequent anticancer therapy, if any. Participants who die without a reported prior progression per Investigator Assessment will be considered to have progressed on the date of death. Participants who did not have any baseline or post baseline tumor assessments and did not die (or died after initiation of the subsequent anti-cancer therapy) will be censored at the randomization date.
Time Frame: From randomization up to the date of the first documented progression (up to approximately 44 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Months | 13.77 [11.53 to 15.70] | 12.19 [10.25 to 14.06]
Statistical Analysis 1: Comparison: Arm A: NIV+mFOLFOX+BEV vs Arm B: mFOLFOX+BEV; Hazard Ratio is Arm A: NIV+mFOLFOX+BEV over Arm B: mFOLFOX+BEV; Test type: Superiority; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.54 to 1.19] — Stratified Cox proportional hazard model

3. Secondary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR)
Description: ORR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). BOR is defined as the best response designation as determined by BICR per RECIST 1.1, recorded between the date of randomization and the date of objectively documented progression per RECIST 1.1 or the date of subsequent anticancer therapy (including tumor-directed radiotherapy and tumor-directed surgery), whichever occurs first. PR is defined as at least a 30% decrease in the sum of diameters of target lesions. CR is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm.
Time Frame: From the date of randomization up to the date of objectively documented progression or the date of subsequent anticancer therapy, whichever occurs first (up to approximately 44 months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Percentage of Participants | 60.6 [51.6 to 69.2] | 45.6 [33.5 to 58.1]

4. Secondary Outcome: Objective Response Rate (ORR) Per Investigator Assessment
Description: ORR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). BOR is defined as the best response designation as determined by tumor assessments by the Investigator per RECIST 1.1, recorded between the date of randomization and the date of objectively documented progression per RECIST 1.1 or the date of subsequent anticancer therapy (including tumor-directed radiotherapy and tumor-directed surgery), whichever occurs first. PR is defined as at least a 30% decrease in the sum of diameters of target lesions. CR is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm.
Time Frame: as for outcome 3
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Percentage of participants | 60.6 [51.6 to 69.2] | 52.9 [40.4 to 65.2]

5. Secondary Outcome: Duration of Response (DoR) Per Blinded Independent Central Review (BICR)
Description: Duration of objective response (DoR) is defined as the time between the date of first confirmed complete response (CR) or partial response (PR) to the date of the first documented tumor progression as assessed by the BICR based on RECIST 1.1 criteria or death due to any cause, whichever occurs first. PR is defined as at least a 30% decrease in the sum of diameters of target lesions. CR is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm.
Time Frame: From randomization up to the date of the first documented progression (per RECIST 1.1) or death due to any cause, whichever occurs first (up to 44 months)
Population: All randomized participants with a CR or PR that were assessed by BICR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 77 | 31
Months | 12.88 [9.00 to 14.72] | 9.26 [7.49 to 11.30]

6. Secondary Outcome: Duration of Response (DoR) Per Investigator Assessment
Description: Duration of objective response (DoR) is defined as the time between the date of first confirmed complete response (CR) or partial response (PR) to the date of the first documented tumor progression as assessed by the investigator based on RECIST 1.1 criteria or death due to any cause, whichever occurs first. PR is defined as at least a 30% decrease in the sum of diameters of target lesions. CR is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm.
Time Frame: as for outcome 5
Population: All randomized participants with a CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 77 | 36
Months | 12.48 [8.87 to 16.72] | 11.07 [9.43 to 17.31]

7. Secondary Outcome: Time to Objective Response Per Blinded Independent Central Review (BICR)
Description: Time to objective response (TTR) is defined as the time from the randomization date to the date of the first confirmed complete response (CR) or partial response (PR) as assessed by BICR. PR is defined as at least a 30% decrease in the sum of diameters of target lesions. CR is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm. TTR is derived for responders only.
Time Frame: From the randomization date up to the date of the first confirmed CR or PR (up to approximately 44 months)
Population: All randomized participants with a CR or PR
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 77 | 31
Months | 2.83 (1.51) | 2.83 (1.45)

8. Secondary Outcome: Time to Objective Response Per Investigator Assessment
Description: TTR is defined as the time from the randomization date to the date of the first confirmed complete response (CR) or partial response (PR) as assessed by investigator. PR is defined as at least a 30% decrease in the sum of diameters of target lesions. CR is defined as the disappearance of all target lesions and the reduction of any pathological lymph nodes to <10 mm. TTR is derived for responders only.
Time Frame: From the randomization date up to the date of the first confirmed CR or PR (up to 44 months)
Population: All randomized participants with a CR or PR
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 77 | 36
Months | 2.83 (2.51) | 2.83 (1.34)

9. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death. For those without documentation of death, OS will be censored on the last date the participant was known to be alive.
Time Frame: From the date of randomization up to the date of death (up to 44 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Months | 30.52 [25.20 to 39.39] | 31.77 [24.38 to 38.70]

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose to 30 days post last dose (up to 45 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 123 | 62
Participants | 122 | 61

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with any grade of serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE v4.0) to determine safety and tolerability. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose to 30 days post last dose (up to 45 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 123 | 62
Participants | 57 | 20

12. Secondary Outcome: Number of Participants Experiencing Death
Description: The number of participants who died during the treatment period
Time Frame: From first dose up to 6 weeks post last dose (up to 46 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 123 | 62
Participants | 87 | 42

13. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: The number of participants with laboratory abnormalities in specific liver tests based on SI conventional units. ALT = Alanine Aminotransferase AST = Aspartate Aminotransferase ULN = Upper Limit of Normal
Time Frame: From first dose up to 30 days post last dose (up to 45 months)
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Number; unit: Participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 123 | 62
Participants
  ALT OR AST > 3XULN | 16 | 6
  ALT OR AST > 5XULN | 7 | 2
  ALT OR AST > 10XULN | 2 | 0
  ALT OR AST > 20XULN | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 0 | 1
  ALP > 1.5XULN | 39 | 20
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN ONE DAY | 2 | 1
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN 30 DAYS | 2 | 1
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY | 0 | 1
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAYS | 0 | 1

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: The number of participants with laboratory abnormalities in specific thyroid tests based on SI conventional units. TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal
Time Frame: From first dose up to 30 days post last dose (up to 45 months)
Population: All Treated Participants with at Least One On-Treatment TSH measurement
Measure: Number; unit: Participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 123 | 60
Participants
  TSH > ULN | 45 | 23
  TSH > ULN WITH TSH <= ULN AT BASELINE | 37 | 16
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 20 | 2
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 11 | 9
  TSH > ULN WITH FT3/FT4 TEST MISSING | 14 | 12
  TSH < LLN | 25 | 3
  TSH < LLN WITH TSH >= LLN AT BASELINE | 22 | 3
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 13 | 0
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 8 | 2
  TSH < LLN WITH FT3/FT4 TEST MISSING | 4 | 1

15. Secondary Outcome: Disease Control Rate (DCR) Per Blinded Independent Central Review (BICR)
Description: Disease Control Rate (DCR) is defined as the percentage of participants whose Best Overall Response (BOR) is complete response (CR) or partial response (PR) or stable disease (SD). CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD is defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 3
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Percentage of participants | 91.3 [85.0 to 95.6] | 83.8 [72.9 to 91.6]

16. Secondary Outcome: Disease Control Rate (DCR) Per Investigator
Description: as for outcome 15
Time Frame: as for outcome 3
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Percentage of participants | 85.8 [85.0 to 95.6] | 77.9 [66.2 to 87.1]

17. Post Hoc Outcome: Progression Free Survival (PFS) Per Blinded Independent Central Review (BICR) - Extended Collection
Description: PFS is the time from randomization to the date of first documented progression, as determined by BICR, or death due to any cause, whichever occurs first. Baseline tumor assessment is defined as tumor scans prior to or on randomization date. Participants who did not have documented progression and did not die or participants who started any subsequent anti-cancer therapy without a prior reported progression were censored on date of last tumor assessment on or prior to initiation of the subsequent anticancer therapy, if any. Participants who died without prior progression were considered to have progressed on the date of death. Participants who did not have any baseline assessments and did not die (or died after initiation of the subsequent anti-cancer therapy) were censored at the randomization date. Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date.
Time Frame: From randomization to up to the date of the first documented progression (up to 44 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
Number analyzed (Participants) | 127 | 68
Months | 11.99 [9.99 to 15.74] | 12.02 [10.25 to 13.37]
Statistical Analysis 1: Comparison: Arm A: NIV+mFOLFOX+BEV vs Arm B: mFOLFOX+BEV; Hazard Ratio is Arm A: NIV+mFOLFOX+BEV over Arm B: mFOLFOX+BEV; Test type: Superiority; p = 0.5041, Log Rank — Stratified regular log-rank test; Hazard Ratio (HR) = 0.88, 80% CI 2-sided [0.67 to 1.15] — Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm A: NIV+mFOLFOX+BEV vs Arm B: mFOLFOX+BEV; Hazard Ratio is Arm A: NIV+mFOLFOX+BEV over Arm B: mFOLFOX+BEV; Test type: Superiority; p = 0.5041, Log Rank — Stratified regular log-rank test; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.58 to 1.32] — Stratified Cox proportional hazard model

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 58 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 45 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Arm A: NIV+mFOLFOX+BEV | Arm B: mFOLFOX+BEV
All-Cause Mortality (participants affected / at risk) | 89/127 | 47/68
Serious Adverse Events (participants affected / at risk) | 67/123 | 25/62
Other Adverse Events (participants affected / at risk) | 122/123 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: NIV+mFOLFOX+BEV (N=123) | Arm B: mFOLFOX+BEV (N=62)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 9 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal obstruction (Gastrointestinal disorders) | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 2 | 2
Infusion site extravasation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Norovirus infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 1
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Stoma prolapse (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: NIV+mFOLFOX+BEV (N=123) | Arm B: mFOLFOX+BEV (N=62)
Anaemia (Blood and lymphatic system disorders) | 32 | 12
Neutropenia (Blood and lymphatic system disorders) | 45 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 7
Tachycardia (Cardiac disorders) | 7 | 1
Hyperthyroidism (Endocrine disorders) | 7 | 1
Hypothyroidism (Endocrine disorders) | 21 | 1
Abdominal distension (Gastrointestinal disorders) | 7 | 2
Abdominal pain (Gastrointestinal disorders) | 40 | 19
Abdominal pain upper (Gastrointestinal disorders) | 12 | 3
Colitis (Gastrointestinal disorders) | 7 | 1
Constipation (Gastrointestinal disorders) | 52 | 21
Diarrhoea (Gastrointestinal disorders) | 74 | 20
Dry mouth (Gastrointestinal disorders) | 15 | 3
Dyspepsia (Gastrointestinal disorders) | 15 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 5
Haemorrhoids (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 83 | 35
Proctalgia (Gastrointestinal disorders) | 12 | 2
Stomatitis (Gastrointestinal disorders) | 28 | 18
Toothache (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 49 | 13
Asthenia (General disorders) | 22 | 6
Chills (General disorders) | 17 | 1
Fatigue (General disorders) | 73 | 38
Influenza like illness (General disorders) | 10 | 1
Malaise (General disorders) | 7 | 3
Mucosal inflammation (General disorders) | 15 | 12
Non-cardiac chest pain (General disorders) | 5 | 4
Oedema peripheral (General disorders) | 12 | 2
Pain (General disorders) | 8 | 3
Pyrexia (General disorders) | 35 | 10
Temperature intolerance (General disorders) | 32 | 14
Hypersensitivity (Immune system disorders) | 10 | 2
Upper respiratory tract infection (Infections and infestations) | 17 | 6
Urinary tract infection (Infections and infestations) | 14 | 7
Fall (Injury, poisoning and procedural complications) | 11 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 27 | 5
Alanine aminotransferase increased (Investigations) | 19 | 11
Aspartate aminotransferase increased (Investigations) | 27 | 10
Blood alkaline phosphatase increased (Investigations) | 15 | 5
Blood creatinine increased (Investigations) | 11 | 2
Neutrophil count decreased (Investigations) | 39 | 12
Platelet count decreased (Investigations) | 25 | 10
Weight decreased (Investigations) | 18 | 12
White blood cell count decreased (Investigations) | 15 | 5
Decreased appetite (Metabolism and nutrition disorders) | 47 | 16
Dehydration (Metabolism and nutrition disorders) | 26 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 3
Dizziness (Nervous system disorders) | 22 | 9
Dysgeusia (Nervous system disorders) | 25 | 12
Headache (Nervous system disorders) | 25 | 6
Hypoaesthesia (Nervous system disorders) | 4 | 6
Neuropathy peripheral (Nervous system disorders) | 54 | 21
Neurotoxicity (Nervous system disorders) | 12 | 2
Paraesthesia (Nervous system disorders) | 11 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 45 | 28
Taste disorder (Nervous system disorders) | 8 | 2
Anxiety (Psychiatric disorders) | 13 | 2
Depression (Psychiatric disorders) | 13 | 3
Insomnia (Psychiatric disorders) | 33 | 10
Proteinuria (Renal and urinary disorders) | 18 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 2
Rash (Skin and subcutaneous tissue disorders) | 14 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9 | 4
Hypertension (Vascular disorders) | 40 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03414983/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03414983/SAP_001.pdf